CLINICAL TRIAL: NCT01279525
Title: EFFECTIVENESS OF A MULTIFACTORIAL INTERVENTION PROGRAM TO REDUCE FALLS INCIDENCE AMONG COMMUNITY-LIVING ELDERLY PEOPLE
Brief Title: Intervention to Reduce Falls Incidence
Acronym: EPICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andalusian Regional Ministry of Health (Other Government)
Collaborators: Andalusian Society of Family Medicine (Unknown); Spanish Society of Family and Community Medicine (Other)
Responsible Party: Luis Angel Pérula de Torres, Andalusian Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 279/03; PI-279/03 (Other: Health Department of the Andalusian Region Government)
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Patient Fall
Keywords: Falls; Prevention; Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multifactorial intervention (Experimental): Multifactorial intervention to prevent falls
  Interventions: Device: multifactorial

INTERVENTIONS:
Device: multifactorial — individual advice, information leaflet, physical exercise workshop and home visits

SUMMARY:
The purpose of this study is to determine the effectiveness of a multifactorial intervention program to prevent falls among the elderly as compared to a brief intervention.

DETAILED DESCRIPTION:
The objective of this research is to verify if a simple multifactorial intervention program that is applicable in PC settings is more effective to decrease fall incidence than a brief advice for community-living people aged 70 or older.

ELIGIBILITY:
Inclusion Criteria:

* Patients residing in the community

Exclusion Criteria:

* to be institutionalized
* Immobilized or bedridden
* Present a terminal disease or severe psychiatric illness
* Have contraindications to physical exercise

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 404 (Actual)
Dates: Start 2005-01; Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
fall incidence rate

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Pérula, Ph D, Principal Investigator — Andalusian Health Service
Locations (1):
- Unidad Docente de Medicina Familiar y Comunitaria, Córdoba, Cordoba, Spain

REFERENCES:
- [Derived] Perula LA, Varas-Fabra F, Rodriguez V, Ruiz-Moral R, Fernandez JA, Gonzalez J, Perula CJ, Roldan AM, de Dios C; EPICA Study Collaborative Group. Effectiveness of a multifactorial intervention program to reduce falls incidence among community-living older adults: a randomized controlled trial. Arch Phys Med Rehabil. 2012 Oct;93(10):1677-84. doi: 10.1016/j.apmr.2012.03.035. Epub 2012 May 15. PMID 22609117